CLINICAL TRIAL: NCT06934044
Title: A Phase Ib, Open-Label, Single-Arm, Multicenter Trial Evaluating the Pharmacokinetics, Safety, and Efficacy of Cevostamab in Chinese Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study Evaluating the Pharmacokinetics, Safety, and Efficacy of Cevostamab in Chinese Participants With Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YO43835
Record Dates: First submitted 2025-04-09; First posted 2025-04-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cevostamab (Experimental): Participants will receive cevostamab administered by intravenous (IV) infusion in 21-day cycles.
  Interventions: Drug: Cevostamab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Cevostamab — Cevostamab will be administered intravenously on a 21-day cycle.
Drug: Tocilizumab — Tocilizumab will be administered for the treatment of cytokine release syndrome (CRS) when necessary.

SUMMARY:
This study will evaluate the pharmacokinetics (PK), safety, and efficacy of cevostamab in participants with relapsed or refractory (R/R) multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of MM based on standard International Myeloma Working Group (IMWG) criteria
* Evidence of progressive disease based on investigators determination of response by IMWG criteria on or after their last dosing regimen
* Current relapsed or refractory (R/R) disease status
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* Agreement to protocol-specified assessments, including bone marrow biopsy and aspirate samples as detailed in the protocol
* Resolution of AEs from prior anti-cancer therapy to Grade =< 1 or better
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception during the treatment period and for at least 5 months after the final dose of cevostamab and for 3 months after the last dose of tocilizumab was administered
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agree to refrain from donating sperm during the treatment period and for at least 2 months after the final dose of tocilizumab (if applicable) to avoid exposing the embryo

Exclusion Criteria:

* Unable to comply with protocol-mandated hospitalization
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 5 months after the final dose of cevostamab or tocilizumab or within 3 months after the last dose of tocilizumab (if applicable)
* Prior treatment with cevostamab or another agent with the same target
* Prior use of any monoclonal antibody (mAb), radioimmunoconjugate, or ADC as anti-cancer therapy within 4 weeks before first study treatment, except for the use of non-myeloma therapy
* Prior treatment with systemic immunotherapeutic agents, including but not limited to, cytokine therapy and anti-CTLA-4, anti-PD-1, and anti-PD-L1
* Prior treatment with CAR-T cell therapy within 12 weeks before first cevostamab infusion
* Known treatment-related, immune-mediated adverse events associated with prior checkpoint inhibitors
* Treatment with radiotherapy, any chemotherapeutic agent, or treatment with any other anti-cancer agent within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to first study treatment
* Autologous stem cell transplantation (SCT) within 100 days prior to first study treatment
* Prior allogeneic SCT
* Prior solid organ transplantation
* History of autoimmune disease
* History of confirmed progressive multifocal leukoencephalopathy
* History of severe allergic or anaphylactic reactions to mAb therapy
* Known history of amyloidosis
* Lesions in proximity of vital organs that may develop sudden decompensation/deterioration in the setting of a tumor flare
* History of other malignancy within 2 years prior to screening, except those with negligible risk of metastasis or death, such as ductal carcinoma in situ not requiring chemotherapy, appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, low-grade, localized prostate cancer not requiring treatment or appropriately treated Stage I uterine cancer
* Current or past history of central nervous system (CNS) disease, such as stroke, epilepsy, CNS vasculitis, neurodegenerative disease, or CNS involvement by MM
* Significant cardiovascular disease that may limit a potential participant's ability to adequately respond to a cytokine release syndrome (CRS) event
* Symptomatic active pulmonary disease or requiring supplemental oxygen
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection at study enrollment, or any major episode of infection requiring treatment with IV (intravenous) antimicrobials where the last dose of IV antimicrobial was given within 14 days prior to first study treatment
* Active symptomatic COVID-19 infection at study enrollment or requiring treatment with IV antiviral where the last dose of IV antiviral treatment was given within 14 days prior to first study treatment.
* Positive and quantifiable Epstein-Barr virus (EBV) polymerase chain reaction (PCR) or cytomegalovirus (CMV) PCR prior to first study treatment
* Known or suspected chronic active EBV infection
* Known history of hemophagocytic lymphohistiocytosis (HLH) or macrophage activation syndrome (MAS)
* Known history of Grade >=3 CRS or immune effector cell-associated neurotoxicity syndrome (ICANS) with prior bispecific therapies
* Recent major surgery within 4 weeks prior to first study treatment
* Positive serologic or PCR test results for acute or chronic hepatitis B virus (HBV) infection
* Acute or chronic hepatitis C virus (HCV) infection
* Known history of human immunodeficiency virus (HIV) seropositivity
* Administration of a live, attenuated vaccine within 4 weeks before first study treatment or anticipation that such a live attenuated vaccine will be required during the study
* Treatment with systemic immunosuppressive medications, with the exception of corticosteroid treatment <= 10 mg/day prednisone or equivalent, within 2 weeks prior to first study treatment
* History of illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Any medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2028-05-08 (Estimated); Study Completion 2028-05-08 (Estimated)

PRIMARY OUTCOMES:
Serum Concentration of Cevostamab at Specified Timepoints | Cycle 1 Day 1 (C1D1) up to approximately 2 years. Each cycle=21 days
Percentage of Participants with Adverse Events | Baseline up to approximately 2 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline up to approximately 2 years
Rate of Complete Response (CR) or Better | Baseline up to approximately 2 years
Rate of Very Good Partial Response (VGPR) or Better | Baseline up to approximately 2 years
Duration of Response (DOR) | Baseline up to approximately 2 years
Progression-free Survival (PFS) | Start of study treatment to first date of disease progression, relapse or death from any cause, whichever occurs first (up to approximately 2 years)
Time to First Response (for Participants who Achieve a Response of Partial Response (PR) or Better) | Baseline up to approximately 2 years
Time to Best Response (for Participants who Achieve a Response of PR or Better) | Baseline up to approximately 2 years
Overall Survival (OS) | Baseline up until death from any cause (up to approximately 2 years)
Minimal Residual Disease (MRD) Negativity (for Participants who Achieve a Response of CR or Better) | Baseline up to approximately 2 years
MRD Negativity (for all Efficacy-evaluable Participants) | Baseline up to approximately 2 years
Number of Anti-drug Antibody (ADAs) Against Cevostamab at Baseline | Baseline
Percentage of Participants with ADAs Against Cevostamab During the Study | Up to approximately 2 years
Number of Participants Reporting Presence, Frequency, Severity, and/or Degree of Interference with Daily Function of Symptomatic Treatment Toxicities Assessed by NCI Patient-Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to approximately 2 years
Number of Participants Reporting Each Response Option for Treatment Side-effect Bother Single-item General Population, Question 5 (GP5) from the Functional Assessment of Cancer Therapy-General Questionnaire; (FACT-G) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- China (5):
  - Sun yat-sen University Cancer Center, Guangzhou, Guangdong
  - Tianjin Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No